CLINICAL TRIAL: NCT01518400
Title: A Research Database for Survivors of Childhood Cancer
Brief Title: LIFE Cancer Survivorship Database for Pediatric Cancer
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, David Freyer, DO, MS, Director, LIFE Cancer Survivorship and Transition Program, Children's Hospital Los Angeles
Other Study IDs: CCI-09-00027
Record Dates: First submitted 2012-01-11; First posted 2012-01-26 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2021-08

CONDITIONS: Pediatric Cancer
Keywords: Pediatric Cancer; Cancer Late Effects; Cancer Survivor; Cancer Survivorship
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eligible Population: Cancer Survivors of all ages (Must be diagnosed with cancer at 21 years or younger)

SUMMARY:
The purpose of this study is to develop a mechanism for utilizing the comprehensive clinical database of childhood cancer survivors at Childrens Hospital Los Angeles (CHLA) for research purposes. Using clinical information obtained from follow-up visits of childhood cancer survivors, the database will focus on interventions to improve health status and health-related quality of life in childhood cancer survivors. This study allows for establishment and analyses of a research database for LIFE survivors by the investigators listed herein. Over the last three decades, there has been marked improvement in survival following childhood cancer, with 5-year survival rates now approaching 80%. However, the use of cancer therapy at an early age can result in complications that may not be apparent until years later as the child matures. These resulting complications, called late effects, are principally related to the specific therapy employed and the age of the child at the time the therapy was administered. Late effects may affect virtually every body system and substantially impair quality of life. As many as two-thirds of childhood cancer survivors develop at least one late effect as a result of treatment, and approximately one-third have a late effect classified as severe or life threatening.

DETAILED DESCRIPTION:
Eligibility Criteria: Eligibility criteria include (1) a history of cancer or similar illness diagnosed before 22 years of age; (2) cancer in remission. Methods: For subjects enrolled on this study, clinical data will be entered into the LIFE database as routinely done for all survivors, but tagged so that research analyses may be carried out and limited only to those who are enrolled on this study.

ELIGIBILITY:
Inclusion Criteria:

1. Been diagnosed with cancer or similar disease
2. Been diagnosed with cancer at 21 years of age or younger
3. Be currently off treatment and disease free

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population diagnosed with cancer at 21 years of age or younger
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2009-02; Primary Completion 2050-01 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
create a database of Cancer Survivors | Annual (up to 40 years)
  To use the information gained from this assessment for identification of risk factors and populations at risk, and to develop interventions to improve health status and quality of life (QOL) in childhood cancer survivors.

CONTACTS AND LOCATIONS:
Overall Officials: David Freyer, DO, MS, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- See also: LIFE Cancer Survivorship Clinic — http://chla.org/LIFE